CLINICAL TRIAL: NCT00947635
Title: Cholesterol and Fatty Acid Synthesis in Islet and Liver Transplant Patients and Effect of Dietary Intervention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Michael T. Clandinin, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Islet-Liver-MTC
Record Dates: First submitted 2009-07-22; First posted 2009-07-28 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2009-07

CONDITIONS: Immunosuppression; Hyperlipidemias; Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes; Transplants; Immunosuppression; Hyperlipidemia; Nutrition Therapy
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Islet transplant (Experimental): People with Type 1 diabetes undergoing islet transplantation
  Interventions: Dietary Supplement: Dietary intervention - supplements
- Liver transplant (Experimental): People with liver failure undergoing liver transplantation
  Interventions: Dietary Supplement: Dietary intervention - supplements
- Control (Experimental): Healthy normal people which serve as control group
  Interventions: Dietary Supplement: Dietary intervention - supplements

INTERVENTIONS:
Dietary Supplement: Dietary intervention - supplements — Supplement bar & spread formulated with key nutrients (fish oil, phytosterols, almonds, soy protein) shown to help in reducing blood lipid levels

SUMMARY:
The purpose is to investigate possible mechanisms of increased blood lipid levels following transplantation, and also to see if a comprehensive dietary intervention is effective in reducing blood lipid levels in post-transplant patients.

DETAILED DESCRIPTION:
Post-transplantation patients frequently have an increase in blood lipid levels presumed to be due to immunosuppressive agents, however it is currently unknown the mechanisms by which this occurs. Dietary interventions have frequently been unsuccessful in these patients, which may be due to single-nutrient interventions and lack of support and guidance. This research will use stable isotope methods to estimate cholesterol and fatty acid synthesis to determine if these pathways are affected by immunosuppression in patients before and after islet and liver transplant. In addition, it will be determined if a multi-nutrient dietary intervention will be implemented post-transplant can reduce blood lipid levels in to prevent further polypharmacy these patients.

ELIGIBILITY:
Inclusion Criteria:

* on islet or liver transplant list
* post-transplant >3 months
* physically able to participate in study and intervention

Exclusion Criteria:

* < 18 years of age
* family history of premature cardiovascular disease or familial hyperlipidemia (control subjects)
* cholestatic diseases (liver transplant patients)
* type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cholesterol and fatty acid synthesis | Pre-transplant, post-transplant (>3 months after transplant, up to 2 years) and post-dietary intervention (1 month after post-transplant measurement)

SECONDARY OUTCOMES:
Blood lipid levels | Pre-transplant, post-transplant (>3 months after transplant, up to 2 years) and post-dietary intervention (1 month after post-transplant measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Clandinin, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada